CLINICAL TRIAL: NCT05655338
Title: Antimicrobial Photodynamic Therapy in Treatment of Aggressive Periodontitis (Stage III, Grade C Periodontitis): A Comparison Between Photodynamic Therapy and Antibiotic Therapy as an Adjunct to Non-Surgical Periodontal Treatment
Brief Title: Antimicrobial Photodynamic Therapy in Treatment of Aggressive Periodontitis (Stage III, Grade C Periodontitis)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ljubljana (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PHOTODYNAMICTHERAPY
Record Dates: First submitted 2022-11-23; First posted 2022-12-19 (Actual); Last update posted 2022-12-19 (Actual); Status verified 2022-12

CONDITIONS: Aggressive Periodontitis
Keywords: Photodynamic therapy; Antibiotic therapy
MeSH Terms: conditions — Aggressive Periodontitis | interventions — Amoxicillin; Metronidazole

STUDY DESIGN:
Who Masked: Care Provider
Masking Description: The blindness of the examiner was ensured by restriction of access to the patients' data. Only the supervisor (MP) had access to the allocation data and therefore knew which patients received additional aPDT treatment.
  Periodontal examinations of 5 randomly selected individuals were carried out twice by the same examiner, and the second measurements were repeated after two weeks. The reproducibility of assessing all periodontal parameters was tested. Intra-examiner calibration scores were 0.95.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ANTIMICROBIAL PHOTODYNAMIC THERAPY (Experimental): The patients received antimicrobial photodynamic therapy after non-surgical periodontal treatment
  Interventions: Device: antimicrobial photodynamic therapy
- SYSTEMIC ANTIBIOTICS (Experimental): The patients received systemic antibiotics after non-surgical periodontal treatment
  Interventions: Drug: systemic antibiotics

INTERVENTIONS:
Device: antimicrobial photodynamic therapy
  Other Names: HELBO TheraLite Laser
  Arms: ANTIMICROBIAL PHOTODYNAMIC THERAPY
Drug: systemic antibiotics
  Other Names: Amoxicillin (Hiconcil); Metronidazole (Efloran)
  Arms: SYSTEMIC ANTIBIOTICS

SUMMARY:
Treatment of aggressive periodontitis (stage III, grade C periodontitis) represents a big challenge. The aim of the study was to compare the long-term results of antimicrobial photodynamic therapy (aPDT) and antibiotic therapy as an adjunct to conventional non-surgical therapy in patients with aggressive periodontitis. Clinical parameters of probing depth, clinical attachment level and bleeding on probing (BOP) were assessed at baseline, 3, 6, 9 and 12 months after treatment.

DETAILED DESCRIPTION:
Background: Treatment of aggressive periodontitis (stage III, grade C periodontitis) represents a big challenge. The aim of the study was to compare the long-term results of antimicrobial photodynamic therapy (aPDT) and antibiotic therapy as an adjunct to conventional non-surgical therapy in patients with aggressive periodontitis. Materials and methods: Twenty subjects with untreated aggressive periodontitis (stage III, grade C periodontitis) were divided into two groups: the test group (TG) received non-surgical therapy and two sessions of aPDT using a laser (HELBO TheraLite laser) with a wavelength of 670nm associated with HELBO Blue photosensitizer, and the control group (CG) received non-surgical therapy and antibiotics (amoxicillin 500mg and metronidazole 400mg, 7 days). Clinical parameters of probing depth, clinical attachment level and bleeding on probing (BOP) were assessed at baseline, 3, 6, 9 and 12 months after treatment.

ELIGIBILITY:
Inclusion Criteria:

* aggressive periodontitis (stage III, grade C periodontitis)
* nonsmokers
* at least 20 teeth in oral cavity
* systemically healthy

Exclusion Criteria:

* any previous periodontal treatment
* smoking
* pregnancy
* ingestion of systemic antibiotics within three months before therapy

Ages: 18 Years to 38 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2015-01-10 (Actual); Primary Completion 2016-06-30 (Actual); Study Completion 2016-06-30 (Actual)

PRIMARY OUTCOMES:
Probing depth reduction | 3 months
  Change in probing depth
Bleeding on probing | 3 months
  Bleeding after measurement of probing depth

SECONDARY OUTCOMES:
Clinical attachment loss | 3 months
  Change in clinical attachment

CONTACTS AND LOCATIONS:
Overall Officials: Boris Gaspirc, Assoc.prof., Study Chair — University of Ljubljana

IPD SHARING:
Plan to Share IPD: No